CLINICAL TRIAL: NCT06016946
Title: Friedreich Ataxia Global Clinical Consortium UNIFIED Natural History Study
Acronym: UNIFAI
Status: Recruiting | Type: Observational
Sponsor: Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: 1016
Record Dates: First submitted 2023-08-18; First posted 2023-08-30 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Friedreich Ataxia
Keywords: Rare Disease; Neuro-degenerative disease; Ataxia; Neurodegenerative Diseases; Neurologic Manifestations; Genetic Diseases, Inborn
MeSH Terms: conditions — Friedreich Ataxia; Rare Diseases; Ataxia; Neurodegenerative Diseases; Neurologic Manifestations; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Biospecimen Retention: Samples With DNA — Whole blood may be collected as a one-time procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is a global, multicenter, prospective, longitudinal, observational natural history study that can be used to understand the disease progression and support the development of safe and effective drugs and biological products for Friedreich ataxia.

DETAILED DESCRIPTION:
The UNIFAI Study: Friedreich Ataxia Global Clinical Consortium UNIFIED Natural History Study is a global research study designed to provide a deep and evolving understanding of the natural history of this rare and debilitating genetic disorder as well as inform clinical trial design and implementation.

Friedreich's Ataxia is a rare, inherited, multi-system condition characterized by progressive neurological and cardiac symptoms. It is caused by mutations in the FXN (frataxin) gene.

The UNIFAI study is a multicenter, prospective, longitudinal, observational study, which means that all data about the natural disease course will be captured at study visits conducted annually according to a single protocol for all sites. This study will recruit participants with FA worldwide, to be assessed annually for up to 25 years. Study participation involves yearly study visits with data collected from medical records and history along with clinical outcome assessments including, neurological exams, timed walking tests, upper limb function measures, and patient-reported quality of life assessments, with the option for sites to collect additional ancillary measures related to speech, vision, fatigue, balance and cognition.

This global study is a harmonization of two well-established, long-standing natural history studies in FA that have provided a framework for further investigation of clinical measures that can quantitatively assess FA: FACOMS (US, Canada, Australia, New Zealand, and India) and EFACTS (European countries). These studies have been conducted in parallel with many similarities in study conduct. Uniting these two existing studies and groups of researchers gives greater power to data previously collected as well as future data. It also continues efforts to expand the network of clinical research centers specializing in FA called the FA-Global Clinical Consortium.

Due to advances in understanding the genetic and cellular dysfunction of FA that lead to symptoms observed in affected individuals, there has been significant growth in the discovery and development of therapeutic approaches, many currently being evaluated in clinical trials and a first approved treatment in the United States in 2023. The UNIFAI study aims to build upon this momentum by focusing on several key objectives.

UNIFAI will assess the natural history of FA by collecting data from diagnosed individuals of all ages and stages of disease progression. The data collected includes demographics, medical history, medications, neurological and functional assessments, cardiac examinations, laboratory studies, and health questionnaires. The study will assess and evaluate clinical outcomes in individuals with FA, such as disease progression, symptom severity, and overall quality of life, by various factors that might influence such outcomes such as genetic mutation, demographics (age, geography), co-existing conditions, medications, or treatments. By tracking outcomes over time, researchers aim to discern patterns, trends, and potential variations in subgroups or in the effectiveness of therapies or interventions across a diverse group of participants.

The UNIFAI study aims to play a pivotal role in identifying clinical milestones and changes in natural history over time as new treatments emerge. The study will monitor how these interventions alter the trajectory of the disease, potentially leading to the identification of crucial tipping points, disease landmarks, or stages where interventions can be most impactful. This study has the potential to significantly improve our understanding of FA and lead to more effective treatments and improved outcomes for those living with FA.

The study aims to inform clinical trial design and the development and validation of novel clinical outcome assessments and biomarkers that can be used in clinical trials. The UNIFAI study aims to capture data from a wide and diverse cohort of individuals with FA so that this dataset can be used to inform the selection of inclusion and exclusion criteria and power calculations for trial designs with specific clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Both males and females of any age
2. Individuals with Friedreich ataxia (FA): Participants that meet genetically confirmed diagnosis of Friedreich ataxia
3. Written informed consent provided

   1. Informed consent must be obtained for all participants
   2. For underage participants, they and the parent/ legally authorized representative have to sign the informed consent form, child assent (if applicable)
   3. Persons who are not legally competent require the informed consent of their legally authorized representative

   Exclusion Criteria:
4. Unable or unwilling to provide informed consent
5. Acute or ongoing medical or other conditions that would interfere with the conduct and assessments of the study
6. For any reason in the opinion of the investigator, participant would be unlikely or unable to comply with study protocol requirements.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will include current participants from the existing FA-COMS and EFACTS natural history studies as well as enroll new individuals with Friedreich ataxia (FA) and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2048-01-28 (Estimated); Study Completion 2048-01-28 (Estimated)

PRIMARY OUTCOMES:
Change in modified Friedreich Ataxia Rating Scale (mFARS) Score | Baseline, Year 1-25
  The modified Friedreich Ataxia Rating Scale (mFARS) is a disease-specific scale that measures progression of neurological effects of FA. The mFARS is a validated and reliable scale; comprised of the neurologic component of the FARS and evaluates bulbar, upper limb, lower limb, and upright stability/gait function. For each item, responses categorize the corresponding neurological finding, and the findings are assigned a score ranging from 0 to 3, 4, or 5 with 0 being normal and higher numbers indicative of greater impairment. The score ranges from 0 to 93. The score will be compared to the previous year annually for up to 25 years.
Change in Scale for the Assessment and Rating of Ataxia (SARA) Score | Baseline, Year 1-25
  The Scale for the Assessment and Rating of Ataxia (SARA) is a semi-quantitative assessment of ataxia, measuring ataxia of upper limb, lower limb, gait, balance and speech. It has eight items: gait, stance, sitting, speech disturbance, finger chase, nose-finger test, fast alternating hand movement, and heel-shin slide. The total score ranges from 0 (no ataxia) to 40 (severe ataxia). The score will be compared to the previous year annually for up to 25 years.
Change in FA Activities of Daily Living (ADL) Score | Baseline, Year 1-25
  The FARS-ADL is a subsection of the FARS questionnaire that assesses activities of daily living, including speech, personal hygiene, feeding, and mobility. Participants rank each category using a scale of 0 (normal) to 4 (severe disability/ inability to carry out activity independently), with lower scores indicative of "normal" function/activity. The score will be compared to the previous year annually for up to 25 years.
Change in Upright Stability (US) Score | Baseline, Year 1-25
  The Upright Stability (US) assessment is part of the neurological examination within the Modified Friedreich Ataxia Rating Scale (mFARS). This component comprises nine items: sitting position, stance with feet apart, stance with feet apart and eyes closed, stance with feet together, stance with feet together and eyes closed, tandem stance, stance with dominant foot, tandem walk, and gait. The score ranges from 0 to 9, with a higher score reflecting poorer upright stability (i.e., greater neurological severity). The score will be compared to the previous year annually for up to 25 years.

SECONDARY OUTCOMES:
Change in 9-hole peg test mean time (seconds) | Baseline, Year 1-25
  The 9 Hole Peg Test (9HPT) examines finger dexterity and involves placing and removing nine pegs in a pegboard in the quickest possible time. Two consecutive trials of the dominant hand, followed immediately by two consecutive trials of the non-dominant hand, are undertaken. The average time in seconds taken to complete the task, for each of the dominant and non-dominant hand, is calculated. The 9HPT has high intra- and inter-rater reliability and is the most commonly used measure of upper limb function in FA. The score will be compared to the previous year annually for up to 25 years.
Change in Timed walk (25-foot or 8-meter) mean time (seconds) | Baseline, Year 1-25
  The timed 25-foot/8-meter walk examines upright stability, balance and mobility and involves walking a predetermined distance. Two consecutive trials are undertaken. The average time in seconds taken to complete the task, is calculated. The score will be compared to the previous year annually for up to 25 years.
Change in Speech analysis scores | Baseline, Year 1-25
  A battery of speech evaluations will be administered and recorded on a laptop for analysis, using Redenlab software. This will include: reading of a phonetically-balanced passage, sustained vowel sound, listing days of the week, repeating syllables, and a monologue task. This will form a measure of dysarthria. Redenlab is a US-Australian speech-testing company, https://redenlab.com. The score will be compared to the previous year annually for up to 25 years.
Change in Ataxia Instrumented Measures (AIMs)clinical severity score | Baseline, Year 1-25
  The Ataxia Instrumented Measures (AIMs) system consists of three components: 1) the data logger which is either a spoon, cup or pendant each containing sensors, Wi-Fi and processor; 2) algorithms that distinguishes between movements made by control and users with ataxia and grades the severity of ataxia when detected; and 3) ataxia scores presented in a manner that has utility for clinicians (the AIM "score"). This score is continuous and features an ataxia severity threshold which has been established through the process of machine learning and is based on the separation between individuals with ataxia and control participants. Any value below the severity threshold of a specific device is expected for controls/very mild ataxia, and any value beyond is expected for individuals with moderate/severe ataxia. The score will be compared to the previous year annually for up to 25 years.
Change in Lower Contrast Letter Acuity test score | Baseline, Year 1-25
  Contrast letter acuity for vision will be assessed using back-lit Low-Contrast Sloan Letter Charts (LCSLCs). Participants will sit at an eye distance of 2 metres from the chart. Binocular vision will be assessed using participants' normal corrective lenses where relevant. Participants are required to read each letter on the chart. Three charts will be presented, with three different visual contrast levels: 100% (equivalent to high-contrast visual acuity), 2.5%, and 1.25%. The maximum total score across the three charts (number of letters read correctly) is 240. Scores for each individual chart will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: David Lynch, MD, Principal Investigator — Children's Hospital of Philadelphia; Jorg B Schulz, Prof, Principal Investigator — University Hospital, Aachen
Locations (34):
- United States (9):
  - UCLA Ataxia Center, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - University of Florida - Neurology, Gainesville, Florida
  - USF Ataxia Research Center, Tampa, Florida
  - Emory University Hospital - Neurology, Atlanta, Georgia
  - University of Iowa, Stead Family Children's Hospital, Iowa City, Iowa
  - Ohio State University - Neurology, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- Murdoch Childrens Research Institute, Parkville, Victoria, Australia
- Medical University Innsbruck, Department of Neurology, Innsbruck, Austria
- Université Libre de Bruxelles, Hôpital Erasme, Dpt of Neurology, Brussels, Belgium
- University of Campinas, Campinas, Brazil
- Canada (3):
  - The Hospital for Sick Children, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Health Centre - Montreal Neurological Institute, Montreal, Quebec
- Motol University Hospital, Centre for Hereditary Ataxias, Prague, Czechia
- France (2):
  - Paris Brain Institute, Paris
  - Hôpital de Hautepierre, Service de Neurologie, Strasbourg
- Germany (4):
  - University Hospital Aachen, Dept. of Neurology, Aachen
  - Deutsches Zentrum Für Neurodegenerative Erkrankungen, Bonn
  - University of Munich, Dept. of Neurology, Friedrich-Baur-Institut, Munich
  - University of Tübingen, Dept. of Neurodegenerative Diseases, Hertie-Institute for Clinical Brain Research, Tübingen
- National and Kapodistrian University of Athens, Neurogenetics Unit, Athens, Greece
- All India Institute of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi, India
- Tallaght University Hospital, Department of Neurology, Dublin, Ireland
- Italy (3):
  - Referente Clinico-Scientifico di Polo IRCCS "E. Medea", Conegliano
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Bambino Gesù Children's Hospital, Department of Neurosciences, Roma
- Stichting Radboud Universitair Medisch Centrum, Nijmegen, Netherlands
- Auckland City Hospital, Auckland, New Zealand
- Spain (2):
  - Hospital Sant Joan de Déu, Servicio de Neurología, Barcelona
  - Hospital Universitario La Paz, Servicio de Neurologia, Madrid
- University College of London, Ataxia Centre, National Hospital for Neurology and Neurosurgery, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided